CLINICAL TRIAL: NCT02769013
Title: Assessing the Effect of Neglected Tropical Diseases on Plasmodium Falciparum Transmission in an Area of Co-endemicity
Acronym: TRANSMAL
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Transmal study version 2.0
Record Dates: First submitted 2016-04-21; First posted 2016-05-11 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2017-10

CONDITIONS: Malaria Transmission
Keywords: Schistosoma haematobium plasmodium falciparum transmission

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample and urine collection potentially containing genetic material of Plasmodium falciparum and Schistosoma haematobium
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- S. haematobium positives in Gabon: Asymptomatic volunteers infected with S. haematobium and living in Gabon
  Interventions: Other: Pre-treatment follow up; Other: S. haematobium treatment; Other: Post treatment follow up; Other: Olfactometer experiment
- S. haematobium negatives in Gabon: Volunteers not infected with S. haematobium and living in Gabon
  Interventions: Other: Pre-treatment follow up; Other: Post treatment follow up; Other: Olfactometer experiment
- S. haematobium positives in Ghana: Asymptomatic volunteers infected with S. haematobium and living in Ghana
  Interventions: Other: Pre-treatment follow up; Other: S. haematobium treatment; Other: Post treatment follow up; Other: Olfactometer experiment
- S. haematobium negatives in Ghana: Volunteers not infected with S. haematobium and living in Ghana
  Interventions: Other: Pre-treatment follow up; Other: Post treatment follow up; Other: Olfactometer experiment

INTERVENTIONS:
Other: Pre-treatment follow up — No active intervention; medical support provided if needed
Other: S. haematobium treatment — Praziquantel-treatment for S. haematobium positive volunteers
  Other Names: Praziquantel-treatment
  Groups: S. haematobium positives in Gabon; S. haematobium positives in Ghana
Other: Post treatment follow up — No active intervention; medical support provided if needed.
Other: Olfactometer experiment — No active intervention; medical support provided if needed.

SUMMARY:
Assessing the effect of neglected tropical diseases on Plasmodium falciparum transmission in an area of co endemicity.

DETAILED DESCRIPTION:
The project is divided in three different work packages that cover the life cycle of P. falciparum :

1. In Work Package 1 (WP1) the investigators will assess whether S. haematobium infection increases the human reservoir of P. falciparum by increasing the carriage rate and incidence of P. falciparum gametocytaemia as well as by increasing the proportion and incidence of subject with sub-microscopic P. falciparum infection. The investigators will also determine whether this increase in gametocyte carriage is a consequence of an impairment of the immune response of helminth infected subjects to P. falciparum.
2. In Work Package 2 (WP2) the investigators will determine whether the transmission of the sexual forms of P. falciparum from the human host to mosquito is increased in S. haematobium infected subjects compared to uninfected controls. Moreover the investigators will study whether the immunological changes induced in S. haematobium infected subjects lead to a decrease of the transmission reducing activity of IgG specific to Pfs48/45 and Pfs230 (both capable of blocking/impairing further development of P. falciparum in the mosquito gut).
3. Finally in Work Package 3 (WP3) the investigators will assess whether S. haematobium infection affects the transmission of P. falciparum from the mosquito to the human host. This effect will be determined indirectly by assessing whether S. haematobium infected subjects are more attractive to mosquitoes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged from 6 to 30 years
* Without severe or moderate disease
* Agreement to be enrolled in the study (written informed consent or consent by the legal representative and assent)
* Living in the study area for at least 1 year

Exclusion Criteria:

* Anaemia with haemoglobin less than 8g/dl
* Know sickle cell disease
* Macroscopic haematuria
* Any other know severe disease

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population are subjects aged from 6 to 30 years since both adults and children have been shown to be a reservoir of P. falciparum. Participants will be recruited in two African villages located in Gabon (lambarene) and Ghana Asokwa submetropolitan area in Kumasi, Ghana. Settings in the two locations are different and represent a rural area with very high infectious pressure from helminths infection (S. haematobium and geohelminths) as well as year-round transmission of malaria in the Central African rain forest (Lambaréné) and a more densely populated area in West Africa with pronounced seasonal variation in malaria transmission and high endemicity of S. haematobium but very little other helminthiases due to well-implemented mass treatment campaigns.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Plasmodium falciparum gametocytes and/or asexual blood stages | 15 months
  Presence of Plasmodium falciparum gametocytes and/or asexual blood stages will be assessed by a quantitative real-time PCR assay in the blood obtained from participants. Unit of measurements for both parameters is numbers/µl.

SECONDARY OUTCOMES:
Number of participants with positive serum antibodies specific to the asexual and gametocyte stages of Plasmodium falciparum. | 15 months
  Number of participants with serum antibodies against P. falciparum gametocyte and/or asexual blood stage antigens will be assessed.
Percentage of mosquitoes attracted to Schistosoma-infected participants to non-infected individuals in a wind-tunnel assay. | 15 months
  100 mosquitoes will be released to Schistosoma infected and non-infected participants simultaneously lying in different tents in a two-way olfactometer.

OTHER OUTCOMES:
Proportion of Plasmodium infected Anopheles mosquitoes per individual per night | 3 months
  Mosquitoes will be collected by Human Landing catches and species of mosquitoes and presence of Plasmodium falciparum will be determined by morphology and PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Ulysse ATEBA NGOA, Dr., Principal Investigator — CERMEL, Lambarene, GABON; Oumou MAIGA, PhD, Principal Investigator — KCCR, Kumasi, Ghana
Locations (2):
- Ayôla Akim ADEGNIKA, Lambaréné, Albert Schweitzer Hospital, Gabon
- KCCR, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edoa JR, Adegbite BR, Honkpehedji YJ, Zinsou JF, Boussougou-Sambe ST, Woldearegai TG, Mordmuller B, Adegnika AA, Dejon-Agobe JC. Epidemiology of soil-transmitted helminth infections and the differential effect of treatment on the distribution of helminth species in rural areas of Gabon. Trop Med Health. 2024 Jan 2;52(1):3. doi: 10.1186/s41182-023-00567-z. PMID 38163912
- [Derived] Dejon-Agobe JC, Edoa JR, Honkpehedji YJ, Zinsou JF, Adegbite BR, Ngwese MM, Mangaboula A, Lell B, Woldearegai TG, Grobusch MP, Mordmuller B, Adegnika AA. Schistosoma haematobium infection morbidity, praziquantel effectiveness and reinfection rate among children and young adults in Gabon. Parasit Vectors. 2019 Dec 10;12(1):577. doi: 10.1186/s13071-019-3836-6. PMID 31823806